CLINICAL TRIAL: NCT06673823
Title: Effects Of Lower Extremity Mirror Therapy On Gait Parameters In Children With Hemiplegic Cerebral Palsy.
Brief Title: Effects of Mirror Therapy on Lower Extremity in CP Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR/AHA/24/sharmeen arif
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
Keywords: lower limb, mirror therapy, conventional therapy, spastic CP
MeSH Terms: conditions — Cerebral Palsy | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be conducted to investigate the effects of mirror therapy in children with hemiplegic cerebral palsy. Children in the control group will receive conventional therapy for 60 minutes, while Children in the experimental group will receive 30 minutes of mirror therapy and 30 minutes of conventional therapy, for 12 weeks, 3 days every week
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In the Experimental Group, Mirror Therapy will be applied by covering any birthmarks or scars on the less affected lower extremity (LE) if they obstruct the child's view. The therapy will take place in a distraction-free environment to help each child maintain focus and concentration. A mirror, at least 35 × 25 inches in size, will be placed between both LEs, with the more affected LE concealed behind a black curtain, allowing a clear reflection of the less affected LE. The child will be instructed to observe the mirror image of their more affected LE for one to two minutes. To begin, the therapist will visually demonstrate the technique.
  Interventions: Device: Mirror therapy
- Control group (Active Comparator): In the Control Group, conventional therapy will include exercises such as stride standing to allow weight shifting between extremities, single leg standing, stooping and recovering from a standing position, standing on a balance board, and various balance training exercises. Additionally, the program will incorporate stretching exercises for the hip flexors, adductors, hamstrings, and calf muscles, along with gait training exercises conducted in an open environment.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Device: Mirror therapy — Mirror Therapy (MT) is a non-invasive treatment method aimed at addressing unilateral conditions impacting either the upper or lower limbs. This technique involves placing a mirror along the patient's sagittal plane, allowing the reflection of the unaffected limb to visually overlay the affected limb.
  Arms: Experimental group
Other: conventional therapy — conventional therapy
  Arms: Control group

SUMMARY:
A non-progressive condition that harms the developing brain both during and after birth is cerebral palsy (CP). It is a multifaceted syndrome marked by abnormalities in movement and posture, along with concomitant sensory-motor, cognitive, and behavioral impairments and seizures. CP can be divided into three types based on neurological classification: spastic, athetoid, and ataxic, impairments in motor skills and posture are hallmarks of cerebral palsy. Various strategies have been employed in motor skill improvement interventions. One of them, mirror-mediated treatment, works by stimulating mirror neurons in a specific region of the brain cortex. Mirror-mediated therapy involves the patient observing movement of his or her own limb reflected in a mirror, which activates mirror neurons. The application of mirror treatment improved gait capacity by elevating physical perception and balance ability. The purpose of the study will be to evaluate the effects of mirror therapy in lower limb hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted to investigate the effects of mirror therapy in children with hemiplegic cerebral palsy. Data will be collected at the National Institute of Rehabilitation Medicine in Islamabad following ethical clearance. 26 patients will be enrolled in the study based on inclusion criteria. Patients will be randomly assigned into 2 equal groups for the study. Children in the control group will receive conventional therapy for 60 minutes, while Children in the experimental group will receive 30 minutes of mirror therapy and 30 minutes of conventional therapy, for 12 weeks, 3 days every week. The primary outcome will be measured by Selective Control Assessment of Lower Extremity scale (SCALE), while the secondary outcome will be measured by the Pediatric Balance Scale (PBS). All gait parameters (stride length, step length, step width, cadence and foot angle) will be measured before and after the application of intervention. Data will be analyzed using SPSS 27.0.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years.
* Motor tone of effected lower extremity is 1 to 2 according to modified Ashworth scale.
* Patient with enough cognition to understand and follow instructions

Exclusion Criteria:

* Patients with any other neurological illness affecting their lower extremities (e.g., MS, Parkinson's, peripheral neuropathy).
* Patients with prior fractures of the lower limb (ankle or foot).
* Patients with other forms of musculoskeletal diseases such as severe arthritis, ankle surgery, leg length difference.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Selective Control Assessment of Lower Extremity scale (SCALE): | 12 weeks
  The Selective Control Assessment of the Lower Extremity (SCALE) is a clinical tool used to measure motor control in individuals with cerebral palsy. In this assessment, participants perform specific isolated movements at each joint, and each joint is scored to produce a total score per limb, with a maximum of 10 points per limb. SCALE demonstrates high interrater reliability, with intraclass correlation coefficients between 0.88 and 0.915. The assessment requires minimal training and takes approximately 10 to 15 minutes to complete.
Pediatric Balance Scale (PBS); | 12 weeks
  The Pediatric Balance Scale is an adaptation of the Berg Balance Scale, designed to evaluate functional balance skills in children. It includes 14 items, each scored from 0 (indicating lowest function) to 4 (indicating highest function), with a maximum possible score of 56 points.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmeen Arif, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morris C. Definition and classification of cerebral palsy: a historical perspective. Dev Med Child Neurol Suppl. 2007 Feb;109:3-7. doi: 10.1111/j.1469-8749.2007.tb12609.x. PMID 17370476